CLINICAL TRIAL: NCT02059694
Title: The Application of Recombinant Human Hyaluronidase is Effective for the Use of Local Blocks for Eyelid Surgery
Brief Title: Use of Recombinant Hyaluronidase Human is Effective for the Use of Local Blocks for Eyelid's Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00051289
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Upper Eyelid Surgery
Keywords: Eyelid surgery; local block/anesthesia; hyaluronidase; Bilateral upper eyelid surgery; Duke Eye Centre; Duke Aesthetic Center
MeSH Terms: interventions — Hyaluronoglucosaminidase; Indicator Dilution Techniques; Dental Occlusion; Lidocaine; Epinephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronidase (Experimental): Dilutions (Blocks):
  0.5 mL of lidocaine 2% with epinephrine 1:100,000 and 0.5 mL of marcaine 0.75% and 1 mL (150 U) of rHuPH20 for a total of 75 U/ml
  Interventions: Drug: Hyaluronidase
- Comparitor (Other): 2 mL of lidocaine 2% with epinephrine 1:100,000 without rHuPH20
  Interventions: Other: 2 mL of lidocaine 2% with epinephrine 1:100,000 without rHuPH20

INTERVENTIONS:
Drug: Hyaluronidase
  Other Names: Dilutions (Blocks):; 0.5 mL of lidocaine 2% with epinephrine 1:100,000 and 0.5 mL of marcaine 0.75% and 1 mL (150 U) of rHuPH20 for a total of 75 U/ml
  Arms: Hyaluronidase
Other: 2 mL of lidocaine 2% with epinephrine 1:100,000 without rHuPH20
  Arms: Comparitor

SUMMARY:
To evaluate the use of recombinant hyaluronidase (rHuPH20) as an adjunctive for local anaesthesia, lidocaine 2% with epinephrine 1:100000, for eyelid surgery.

DETAILED DESCRIPTION:
Subjects scheduled for bilateral upper eyelid surgery will be recruited from among the patients of the Duke Eye Center. After consent is obtained following full explanation of the research, subjects will be randomly assigned (1:1 ratio) on the day of the surgery to receive local anaesthesia by either with recombinant hyaluronidase (rHuPH20) or without it. Approximately 2 ml of prepared block will be infiltrated in both upper eyelids.

Dilutions (Blocks):

A) 0.5 mL of lidocaine 2% with epinephrine 1:100,000 and 0.5 mL of marcaine 0.75% and 1 mL (150 U) of rHuPH20 for a total of 75 U/ml B) 2 mL of lidocaine 2% with epinephrine 1:100,000 without rHuPH20

Test preparation will be applied subcutaneously in both upper eyelids by injection using a 30-gauge injection needle with the patient in supine position. Every patient will be injected by the same Oculoplastic surgeon.

A Pinprick pain test will be perform 5 minutes after each injection using a sterile "finger stick" needle at three sites of each upper eyelid. These sites include medial, central and lateral portion of each eyelid, approximately 4 mm above the lid margin. The subject will be asked to rate the degree of pain experienced at each site on a scale from 0 (none) to 10 (severe). An average pain score will be calculated for each eyelid. This will help determine if one of the 2 dilutions have a faster anaesthetic effect.

Patients will also be instructed to inform the surgeon of precisely when the pain began and subsided to accurately record the duration of the pain experienced.

ELIGIBILITY:
* Inclusion Criteria:
* Capable and willing to provide consent
* Has been scheduled for bilateral upper eyelid surgery
* At least 18 years of age
* Exclusion Criteria:
* Unable or unwilling to give consent
* Previous upper eyelid surgery
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Pain sensation | 5 minutes after injection
  Test preparation will be applied subcutaneously in both upper eyelids by injection using a 30-gauge injection needle with the patient in supine position. Every patient will be injected by the same Oculoplastic surgeon.
  A second investigator (masked to the treatment condition of each eye) will test Pinprick pain Sensation 5 minutes after each injection using a sterile "finger stick" needle at three sites of each upper eyelid. These sites include medial, central and lateral portion of each eyelid, approximately 4 mm above the lid margin. The subject will be asked to rate the degree of pain experienced at each site on a scale from 0 (none) to 10 (severe).

SECONDARY OUTCOMES:
Anesthesia duration | After procedure started
  Patients will also be instructed to inform the surgeon of precisely when the pain began and subsided to accurately record the duration of the pain experienced.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Roberts MA, Mendez U, Gilbert RJ, Keim AP, Goldman J. Increased hyaluronan expression at distinct time points in acute lymphedema. Lymphat Res Biol. 2012 Sep;10(3):122-8. doi: 10.1089/lrb.2012.0001. PMID 22984909
- [Background] Rowlett J. Extravasation of contrast media managed with recombinant human hyaluronidase. Am J Emerg Med. 2012 Nov;30(9):2102.e1-3. doi: 10.1016/j.ajem.2012.03.005. Epub 2012 May 23. PMID 22633726
- [Background] Clark LE, Mellette JR Jr. The use of hyaluronidase as an adjunct to surgical procedures. J Dermatol Surg Oncol. 1994 Dec;20(12):842-4. doi: 10.1111/j.1524-4725.1994.tb03718.x. PMID 7798421
- [Background] Wohlrab J, Finke R, Franke WG, Wohlrab A. Efficacy study of hyaluronidase as a diffusion promoter for lidocaine in infiltration analgesia of skin. Plast Reconstr Surg. 2012 Apr;129(4):771e-772e. doi: 10.1097/PRS.0b013e318245ea27. No abstract available. PMID 22456420
- [Background] Kallio H, Paloheimo M, Maunuksela EL. Hyaluronidase as an adjuvant in bupivacaine-lidocaine mixture for retrobulbar/peribulbar block. Anesth Analg. 2000 Oct;91(4):934-7. doi: 10.1097/00000539-200010000-00031. PMID 11004052
- [Background] Nathan N, Benrhaiem M, Lotfi H, Debord J, Rigaud G, Lachatre G, Adenis JP, Feiss P. The role of hyaluronidase on lidocaine and bupivacaine pharmacokinetics after peribulbar blockade. Anesth Analg. 1996 May;82(5):1060-4. doi: 10.1097/00000539-199605000-00032. PMID 8610868